CLINICAL TRIAL: NCT06294418
Title: Non-invasive In-vivo Characterisation of Postoperative Low Grade Gliomas Using Field Cycling Imaging (FCI)
Brief Title: FCI in Post-operative Low Grade Gliomas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Grampian (Other Government)
Collaborators: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1-037-23
Record Dates: First submitted 2024-02-26; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Low grade glioma (Experimental): Patients with postoperative low grade glioma will undergo one FCI scan.
  Interventions: Device: Field Cycling Imaging (FCI)

INTERVENTIONS:
Device: Field Cycling Imaging (FCI) — FCI scan

SUMMARY:
The aim of this pilot study is to explore the utility of a new imaging technique, called Field Cycling Imaging (FCI), in postoperative low grade gliomas.

The main question it aims to answer is if FCI can differentiate subtypes of low grade gliomas. Participants will have one FCI scan.

DETAILED DESCRIPTION:
Standard clinical magnetic resonance imaging (MRI) is the mainstay of diagnosis in brain lesions. It is a powerful imaging technique for the non-invasive investigation of the brain and has been an incredibly successful technology since its commercialisation in the 1980s largely due to its excellent spatial resolution and ability to distinguish multiple tissues in multiple planes. When exogenous contrast agents are used, MRI can demonstrate the breakdown of the blood-brain barrier and provide additional physiological information.

However, standard MRI has limitations in determining the subtypes of tumours, which originate from different cells and therefore contain differing types of proteins. The aim of this project is to establish if there is a difference in the relaxometry (i.e., loss of MRI signal over time) characteristics of different brain lesions using Field Cycling Imaging (FCI), which is a new technology being developed at the University of Aberdeen.

FCI combines the use of a moderately high magnetic field with the ability to probe low magnetic fields so that one can preserve image resolution while also exploiting the high contrast present at low magnetic fields. This provides quantitative data on the molecular dynamics in the tissues, completely non-invasively.

For this study, the research team will use FCI to try to establish if there is a difference in the relaxometry characteristics of different low-grade gliomas. Ten patients with postoperative low grade glioma will be included. Each participant will be asked to undergo one FCI scan only. FCI images will be acquired on dedicated equipment, specifically built for the purpose of imaging human volunteers and patients. Participants will carry on receiving their routine clinical care before and after their scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with post operative low-grade glioma.
* Capacity to give informed consent.
* Capacity to co-operate with the scanning procedures and duration.
* Age 16 and above.
* Participants who can pass through a 50 cm-diameter circular hoop to ensure they will be able to fit inside the scanner.
* Participants who meet the safety criteria for undergoing an MRI scan.
* Participants must be mobile enough to be positioned onto the FCI scanner couch.

Exclusion Criteria:

* MRI-incompatible conditions, as detected in the MRI safety screening form.
* Restrictions to mobility that would prevent the correct positioning in the scanner by trained research radiographer (e.g., severe kyphosis).
* Participants who are unable to give fully informed consent.
* Women who are pregnant.
* Participants who are unable to understand or communicate in English.
* Patients who suffer from claustrophobia.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Differentiation of sub-types of low grade glioma assessed by Field Cycling Imaging (FCI) T1 dispersion profiles | At baseline
  Validation of FCI T1 dispersion profiles as a non-invasive technology to differentiate sub-types of low grade glioma.

CONTACTS AND LOCATIONS:
Overall Officials: Arnab K Rana, Dr, Study Chair — University of Aberdeen
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No